CLINICAL TRIAL: NCT05060926
Title: Intubation Prediction in Sars-CoV-2 Patients Treated With Awake Prone Positioning
Brief Title: Intubation Prediction in COVID-19 Patients Treated With Awake Prone Positioning
Acronym: Intub_prone
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Piquilloud Imboden Lise, Principal Investigator, University of Lausanne Hospitals
Other Study IDs: Intub_prone
Record Dates: First submitted 2021-09-16; First posted 2021-09-29 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2021-09

CONDITIONS: Acute Hypoxemic Respiratory Failure; SARS-CoV-2 Virus
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Awake prone positioning — Awake prone position as long as possible according to the patients' tolerance

SUMMARY:
Retrospective study in Sars-Cov 2 patients hospitalised in ICU. We aim to explore the effects of Awake prone positioning on oxygenation and intubation rate.

ELIGIBILITY:
Inclusion Criteria:

* Sars-CoV-2 pneumonia
* ICU stay
* Severe hypoxemia but non intubated

Exclusion Criteria:

* Intubated before admission
* Denied consent for data analysis
* Do not intubate order at ICU admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sars-CoV-2 pneumonia patients with severe hypoxemia
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Intubation rate | Once between ICU admission and extubation

SECONDARY OUTCOMES:
Alveolo-arterial gradient change | Within 6 hours before and 6 hours after each pronation
Blood gas analysis | Within 6 hours before and 6 hours after each pronation
Respiratory pattern | Within 6 hours before and 6 hours after each pronation
Mortality | Up to 28 days from ICU admission

CONTACTS AND LOCATIONS:
Locations (1):
- Lausanne University Hospitals, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No